CLINICAL TRIAL: NCT07320599
Title: Neuroendoscopic Surgery With Ommaya Reservoir Implantation vs. Burr Hole Drainage for Infantile Postmeningitis Subdural Lesions: Superior Efficacy, Critical Impact of Surgical Timing, and Pathogenic Bacteria as Risk Factors for Progression
Status: Not yet recruiting | Type: Observational
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Wangyikang, Dr, Shengjing Hospital
Other Study IDs: wangyikang@000622
Record Dates: First submitted 2025-09-05; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Meningitis
Keywords: infantile meningitis
MeSH Terms: conditions — Meningitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endoscopic Subdural Fluid Collection Evacuation & Ommaya Reservoir Implantation — Neuroendoscopy offers significant advantages in IPSE/IPSFC management. It enables visualized resection of subdural FIPLs (fibrous cords, purulent debris, septa, most pseudomembranes), improving lesion clearance and reducing pathogen colonization via high-definition visualization. The minimally invasive approach uses a 3-cm incision and 4-6 cm² bone window, minimizing iatrogenic injury to brain and dura. Meanwhile, direct visualization allows exploration of multilocular cavities, septum disruption, and complete drainage, avoiding residual risks of traditional single-burr drainage. Visualized manipulation avoids vessels and functional areas, reducing injury and complications (e.g., epilepsy, deficits), and protecting infant brain development. ORI is crucial in IPSE/IPSFC treatment.

SUMMARY:
Globally, approximately 750,000 cases of infantile meningitis occur annually[1]. Clinical data show infantile postmeningitis subdural fluid collection (IPSFC) is the most common complication of infantile bacterial meningitis (IBM), with a progression rate of 30-60% (39% in standardized treatment cohorts)[2]. Pathogens, predominantly Escherichia coli and Streptococcus pneumoniae, account for 70% of IPSFC cases[3]. IPSFC progresses to subdural empyema (IPSE) in 3.7-17.6% of cases, with 87.1% of IPSE cases occurring in infants <1 year old[4]. Collectively termed infantile postmeningitis subdural space lesions (IPSSL), these conditions impose the highest burden in Sub-Saharan Africa's "Meningitis Belt" and Southeast Asia[5]. IPSE progresses rapidly in infants, with a mortality rate of 18% and 50% of survivors developing neurological sequelae (e.g., epilepsy, motor/intellectual disability, sensory impairment)[6]. While spontaneously resolved IPSFC shows no significant sequelae, prolonged IPSE disrupts brain development, requires extended treatment, and incurs substantial familial burdens.

Causes of IPSFC secondary to IBM include increased subdural capillary permeability (with plasma exudation), cerebrospinal fluid (CSF) circulation/absorption disturbance, immature infantile blood-brain barrier (BBB), and underdeveloped arachnoid granulations[7]. IPSFC typically develops on days 7-10 of IBM and is staged by fluid thickness: Stage I (<0.3 mm), Stage II (3-8 mm), Stage III (>8 mm)[8]. Uncontrolled IBM infection, due to inappropriate antibiotics, inadequate dosage, delayed treatment, or infantile immunocompromise, e.g., preterm infants, allows pathogens to invade and proliferate in the subdural space, inducing local secondary infection, inflammatory cell infiltration, and accumulation of pathogen metabolites/necrotic tissue-ultimately progressing to IPSE[9]. Fibrinogen exudation and fibroblast activation may further form subdural fibrous cords, septa, purulent plaques, inflammatory pseudomembranes, and other fibro-inflammatory proliferative lesions (FIPLs)[10]. IPSE causes more severe mass/toxic effects, requiring aggressive surgical intervention. Cranial MRI shows empyema cavity rim enhancement, heterogeneous internal signals due to fluid collection septa, and dural thickening.

The progression rate of IPSFC to IPSE ranges from 3.7% to 17.6%, influenced by IBM pathogen types, therapeutic intervention, and host immunity[11]. However, large-scale cohort studies on risk factors for this progression remain lacking. Early adequate antibiotic therapy reduces IPSFC incidence by nearly 50%, whereas delayed intervention may accelerate IPSFC onset (day 3-7) via unremitting meningeal permeability[12]. Inadequate antibiotic courses may promote persistent IPSFC progression with FIPLs formation. Some pediatric neurosurgeons advocate extending antibiotic therapy beyond 21 days for IPSFC to prevent progression to IPSE[13].

Despite early antibiotic therapy reducing IBM mortality, IPSSL management remains challenging. A clinical study showed 22.4% of IPSFC cases required surgery, but occult inflammation in infants can prolong IPSFC up to 2 months[14]. Infantile unclosed fontanelles and cranial elasticity increase neurosurgical complication risks. Current consensus suggests asymptomatic/small-volume fluid collections (thickness <5 mm) often resolve spontaneously, obviating intervention[15]. Ultrasound-guided subdural puncture (US-SP-AF) is the first-line invasive treatment, curing about 50% of infants acutely but with a 30-50% recurrence rate. Whether US-SP-AF reduces IPSFC-to-IPSE progression remains controversial. For US-SP-AF-resistant cases, minimally invasive burr hole irrigation (BHID) with silicone tube drainage (3-5 days) is used; BHID shows higher cure rates than US-SP-AF but still has a 20-33% recurrence rate in small cohorts[16].

Neuroendoscopic technique allows rigid endoscope entry into the subdural space for visualized resection of pathological tissues, management of multiloculated cavities, adhesion lysis, and FIPLs irrigation. This approach directly targets the pathological substrate under vision, reducing residual lesions and recurrence rates compared to traditional methods. In adult cohorts, 6-month postoperative fluid collection recurrence rates are only 8% with neuroendoscopy, versus 33% with BHID[17]. However, neuroendoscopic exploration is technically demanding and equipment-dependent. The Ommaya reservoir offers advantages in postoperative management of cerebrospinal fluid-related disorders, including precise drainage, dynamic monitoring of disease progression, and local drug administration. However, it may be prone to catheter obstruction by pathological components[18].

Severe IPSSL causes intracranial hypertension and neurodevelopmental impairment, requiring comprehensive pediatric neurosurgical and pharmacologic strategies. Treatment selection depends on IPSFC/IPSE pathological features. Current stu

ELIGIBILITY:
Inclusion Criteria:

- All enrolled children had received ≥3 weeks of standardized anti-infection therapy, including empirical or susceptibility-guided antibiotics administered intrathecal (post-lumbar puncture) or intravenous and dexamethasone administered intrathecal or intravenous. During conservative management, vital/neurological signs were closely monitored, with regular imaging to assess fluid thickness and empyema progression. Cranial ultrasound (primary modality, ≤3-day intervals) was performed, while CT/MRI were conducted ≤weekly.

Exclusion Criteria:

* subdural fluid collections secondary to viral meningitis; secondary collections with confirmed craniocerebral trauma history; diagnosed tuberculous subdural fluid collection; intracranial space-occupying lesions.

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children undergoing surgical treatment should meet at least one imaging criterion (persistent short-term widening of the subdural space or compression of lateral ventricles; unilateral fluid collection thickness >1 cm for two consecutive weeks; formation of empyema abscess wall or mature empyema) and at least two clinical criteria (head circumference growth rate exceeding normal range or increased fontanelle tension; worsening IPSSL symptoms or persistent poor infection control; manifestations of intracranial hypertension such as repeated vomiting or lethargy; frequent neurological abnormalities like epileptic seizures; asymptomatic cases with fluid/empyema thickness >1 cm for >2 weeks).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
IPSSL-score | 1 year
  This scale incorporates the Hines Neurological Score for Infants (neonatal to 2-year neurofunctional assessment, adapted from traditional Hines Score), intracranial pressure parameters, inflammatory control, and neurological function. The IPSSL-score (total 20 points) shows lower preoperative scores indicate worse symptoms and higher postoperative scores reflect better outcomes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen TM, Chen HY, Hu B, Hu HL, Guo X, Guo LY, Li SY, Liu G. Characteristics of Pediatric Recurrent Bacterial Meningitis in Beijing Children's Hospital, 2006-2019. J Pediatric Infect Dis Soc. 2021 May 28;10(5):635-640. doi: 10.1093/jpids/piaa176. PMID 33491083

DOCUMENTS (2):
  • Study Protocol: _2.0 (2025-12-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT07320599/Prot_000.pdf
  • Study Protocol: _1.0 (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT07320599/Prot_001.pdf